CLINICAL TRIAL: NCT07323485
Title: Effect of Preoperative Inflammatory Biomarkers on Postoperative Delirium in Children Undergoing Circumcision
Brief Title: Inflammatory Biomarkers and Postoperative Delirium in Pediatric Circumcision
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Murat Gul, Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-299
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Delirium; Pediatric Anesthesia; Inflammatory Biomarkers
Keywords: Circumcision; Pediatric Anesthesia; Inflammatory Biomarkers; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of Preoperative Inflammatory Biomarkers — Blood samples will be collected preoperatively to assess inflammatory biomarkers, including the neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), systemic immune-inflammation index (SII), monocyte-to-lymphocyte ratio (MLR), and the systemic inflammation response index (SIRI). These parameters will be analyzed in relation to the incidence of emergence delirium within the first 2 hours following pediatric circumcision.
  No experimental drug or medical device will be used as part of the study; all procedures will be performed within the scope of standard perioperative care.

SUMMARY:
Postoperative delirium may occur in children after general anesthesia, even following short procedures such as circumcision. Preoperative systemic inflammation has been associated with postoperative delirium in adults, but data in pediatric patients are limited. This prospective observational study aims to evaluate the association between preoperative inflammatory biomarkers and postoperative delirium in children aged 2-12 years undergoing elective circumcision under general anesthesia. Inflammatory biomarkers derived from routine complete blood count parameters, including NLR, PLR, MLR, SII, and SIRI, will be analyzed. Postoperative delirium will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale in the post-anesthesia care unit. The relationship between inflammatory biomarkers and delirium development and severity will be evaluated. This study seeks to identify simple preoperative markers that may help predict postoperative delirium risk in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-12 years.
* Patients scheduled to undergo elective circumcision under general anesthesia.
* Patients classified as ASA physical status I-II.
* Patients whose parents or legal guardians provide written informed consent, and whose age-appropriate verbal assent is obtained from the child.
* Patients in whom anesthesia and surgical procedures are performed according to standard institutional protocols throughout the study period.

Exclusion Criteria:

* Children with a history of neurological or psychiatric disorders (e.g., epilepsy, developmental delay, autism spectrum disorder, anxiety disorders).
* Patients classified as ASA physical status III-IV.
* Patients with incomplete preoperative laboratory data or with hematological or hormonal disorders that may affect inflammatory parameters.
* Patients who develop excessive sedation after premedication or whose preoperative assessment cannot be completed.
* Patients with protocol deviations during surgery or anesthesia (e.g., additional medications, prolonged surgical duration, or changes in procedure due to complications).
* Patients whose parents or legal guardians do not provide consent or who decline participation.

Ages: 2 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 2-12 years with ASA physical status I-II undergoing elective circumcision under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Delirium | Within 2 hours postoperatively
  Postoperative delirium will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale.

SECONDARY OUTCOMES:
Correlation between preoperative inflammatory biomarkers (NLR, PLR, SII, SIRI, MLR) and delirium severity (total PAED score). | Within 2 hours postoperatively
  The correlation between preoperative inflammatory biomarkers (NLR, PLR, SII, SIRI, and MLR) and the severity of postoperative delirium, as measured by the total Pediatric Anesthesia Emergence Delirium (PAED) score, will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)